CLINICAL TRIAL: NCT01589432
Title: A Randomized, Double-blind, Placebo and Active-controlled Study of the Electrophysiological Effects of ABT-639 on Spontaneous Activity in C-Nociceptors in Patients With Painful Diabetic Peripheral Neuropathy
Brief Title: A Randomized, Double-blind, Placebo- and Active-controlled Study of the Electric Current Effects of ABT-639 on the Spontaneous Activity of Pain Sensory Receptors in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: M13-383; 2011-005127-40 (EudraCT Number)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Neuropathic Pain
Keywords: Diabetic peripheral neuropathy
MeSH Terms: interventions — 4-chloro-2-fluoro-N-(2-fluorophenyl)-5-(hexahydropyrrolo(1,2-a)pyrazin-2(1H)-ylcarbonyl)benzenesulfonamide; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABT-639 (Experimental)
  Interventions: Drug: ABT-639
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: ABT-639 — two 50 mg oral capsules
  Arms: ABT-639
Drug: Placebo — 2 placebo capsules
  Arms: Placebo
Drug: Lidocaine — 3mg/kg infusion over 30 minutes
  Arms: Lidocaine

SUMMARY:
People with diabetes can, over time develop nerve damage throughout the body with symptoms such as pain, tingling, or numbness (loss of feeling) in the hands, arms, feet and legs.

ELIGIBILITY:
Inclusion Criteria

* Subject is between the ages of 18 to 75 years with a diagnosis of diabetes mellitus and must have a diagnosis of painful distal symmetric diabetic polyneuropathy and presence of ongoing pain due to diabetic peripheral neuropathy for at least 6 months.
* Subject must have an average score of greater than or equal to 4 on the 24 hour average pain score (0-10 numerical rating scale) collected over approximately 7 days prior to the Baseline Visit.

Exclusion Criteria

* Subject has clinically symptomatic neuropathic pain conditions that can not be distinguished from diabetic neuropathic pain or interfere with the pain assessments of diabetic neuropathic pain.
* A subject has newly diagnosed or clinically significant medical conditions or mental disorders that would preclude participation or would interfere with diabetic neuropathic pain assessments or other functions.
* Subject has clinically significant abnormalities in clinical laboratory tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Spontaneous activity in peripheral c-nociceptors | 10 minute intervals over 180 minutes
  Spontaneous activity in peripheral c-nociceptor measured through microneurography

SECONDARY OUTCOMES:
Pain intensity measurements | hourly for 4 hours
  Pain intensity reported on a numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, MD, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 68882, London, United Kingdom

REFERENCES:
- [Derived] Serra J, Duan WR, Locke C, Sola R, Liu W, Nothaft W. Effects of a T-type calcium channel blocker, ABT-639, on spontaneous activity in C-nociceptors in patients with painful diabetic neuropathy: a randomized controlled trial. Pain. 2015 Nov;156(11):2175-2183. doi: 10.1097/j.pain.0000000000000249. PMID 26035253